CLINICAL TRIAL: NCT00619619
Title: Final Report: Multicenter, Open-Label, Safety, Tolerability, And Pharmacokinetic Study To Evaluate Single Ascending Doses And Subsequent Short-Term Administration Of Fixed Doses Of DVS SR Tablets In The Treatment Of Child And Adolescent Outpatients With Major Depressive Disorder
Brief Title: Study Evaluating Desvenlafaxine Succinate Sustained-Release (DVS SR) In The Treatment Of Child And Adolescent Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 3151A6-2000; B2061012; 3151A6-2000-US
Record Dates: First submitted 2008-01-28; First posted 2008-02-21 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Depression; Major Depressive Disorder
Keywords: MDD; Child; Adolescent; Pharmacokinetic; Outpatient; Pediatrics; Depressive Disorder; Major
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release Tablets (DVS SR)

INTERVENTIONS:
Drug: Desvenlafaxine Succinate Sustained-Release Tablets (DVS SR) — DVS SR Tablets of 10mg, 25mg, 50mg, and 100mg. Assigned DVS SR daily doses of 10mg, 25mg, 50mg, 100mg, or 200mg for up to 8 weeks.

SUMMARY:
The primary purpose of this study is to test the safety and tolerability of single ascending doses of Desvenlafaxine Succinate Sustained-Release (DVS SR) in both child and adolescent outpatients with major depressive disorder. This study will also characterize the pharmacokinetic profile of DVS SR in children and adolescents with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatient between 7 and 17 years of age at baseline who meet Diagnostic and Statistic Manual of Mental Disorders, Fourth Edition, Text Revision criteria for major depressive disorder.
* Children's Depression Rating Scale --Revised (CDRS-R) score greater than 40 at the screening and study day -1 (baseline) visits and Clinical Global Impressions Scale--Severity (CGI-S) score of greater than or equal to 4 at the screening and study day -1 (baseline) visits.
* Depression of at least moderate severity with symptoms for at least 1 month before screening and that could, in the investigator's opinion, respond to therapy with antidepressant(s) alone (without concomitant psychotherapy).
* Other inclusion criteria apply.

Exclusion Criteria:

* History or current evidence of a medical condition known to interfere with the absorption or excretion of drugs or a history of surgery known to interfere with the absorption or excretion of drugs; history or presence of any other medical condition that might confound the study or put the study participant at greater risk during participation; known hypersensitivity to venlafaxine.
* History of suicide attempt or gesture in which the intent was suicide or serious self-harm or acute suicidality to such a degree that precaution against suicide must be exercised.
* Current (within 12 months before baseline) psychoactive substance abuse or dependence (including alcohol), manic episode, posttraumatic stress disorder, obsessive-compulsive disorder, or a diagnosis of bipolar disorder or psychotic disorder or current (within 12 months before baseline) generalized anxiety disorder, panic disorder, social anxiety disorder, or attention deficit hyperactivity disorder (ADHD) if considered by the investigator to be primary (causing a higher degree of distress or impairment than MDD) or presence (within 12 months before baseline) of a clinically important personality disorder (such as antisocial, schizotypal, histrionic, borderline, or narcissistic) as assessed during the psychiatric evaluations or history or presence of MDD with psychotic features.
* Other exclusion criteria apply.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2008-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (9):
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, North Miami, Florida
  - Pfizer Investigational Site, Terre Haute, Indiana
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3151A6-2000&StudyName=Study%20Evaluating%20Desvenlafaxine%20Succinate%20Sustained-Release%20%28DVS%20SR%29%20In%20The%20Treatment%20Of%20Child%20And%20Adolescent%20Outpatients%20With%20Major%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment to be given at only 1 dose level at a time for at least the first 6 subjects per dose group. Approximately 6 to 8 subjects were to be enrolled in each of the dose cohorts; 4 dose levels were to be evaluated per age stratum in sequential manner and ascending order (10 to 100 milligrams (mg) for children; 25 to 200 mg for adolescents).
Pre-assignment Details: Screening period 6 to 14 days followed by treatment period (up to 3.5 day inpatient and up to 7.5 week outpatient phase). Participants who enter outpatient period but do not continue into 6-month open-label extension study (NCT00669110) will participate in taper period of 0 to 2 weeks depending on dose of study treatment to which they are assigned.
Groups:
- Desvenlafaxine 10 mg Children: Desvenlafaxine sustained release 10 milligram (mg) tablet
- Desvenlafaxine 25 mg Children; Desvenlafaxine 25 mg Adolescent: Desvenlafaxine sustained release 25 mg tablet on Day 1, 10 mg tablet on Days 4 through 7, 25 mg tablet on Days 8 through 56, 10 mg tablet for 7 day taper.
- Desvenlafaxine 50 mg Children; Desvenlafaxine 50 mg Adolescent: Desvenlafaxine sustained release 50 mg tablet on Day 1, 10 mg tablet on Days 4 through 7, 25 mg tablet on Days 8 through 14, 50 mg tablet on days 15 through 56, 25 mg tablet on taper Days 1 through 7, 10 mg tablet for taper Days 8 through 14.
- Desvenlafaxine 100 mg Children; Desvenlafaxine 100 mg Adolescent: Desvenlafaxine sustained release 100 mg tablet on Day 1, 25 mg tablet on Days 4 through 7, 50 mg tablet on Days 8 through 14, 100 mg tablet on days 15 through 56, 50 mg tablet on taper Days 1 through 7, 25 mg tablet for taper Days 8 through 14.
- Desvenlafaxine 200 mg Adolescent: Desvenlafaxine sustained release two 100 mg tablets on Day 1, 50 mg tablet on Days 4 through 7, 100 mg tablet on Days 8 through 14, two 100 mg tablets on days 15 through 56, 100 mg tablet on taper Days 1 through 7, 50 mg tablet for taper Days 8 through 14.
Period: Overall Study
Arm/Group | Desvenlafaxine 10 mg Children | Desvenlafaxine 25 mg Children | Desvenlafaxine 50 mg Children | Desvenlafaxine 100 mg Children | Desvenlafaxine 25 mg Adolescent | Desvenlafaxine 50 mg Adolescent | Desvenlafaxine 100 mg Adolescent | Desvenlafaxine 200 mg Adolescent
Started | 6 | 7 | 9 | 7 | 7 | 7 | 8 | 8
Entered the Extension Study | 6 (Extension study: 3151A6-2001 (NCT00669110)) | 5 | 8 | 3 | 7 | 6 | 6 | 7
Completed | 6 (Completed=conclusion of Test Article (treatment) phase for all treatment groups in 3151A6-2000.) | 7 | 8 | 6 | 5 | 7 | 7 | 5
Not Completed | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desvenlafaxine 10 mg Children | Desvenlafaxine 25 mg Children | Desvenlafaxine 50 mg Children | Desvenlafaxine 100 mg Children | Desvenlafaxine 25 mg Adolescent | Desvenlafaxine 50 mg Adolescent | Desvenlafaxine 100 mg Adolescent | Desvenlafaxine 200 mg Adolescent | Total
Number analyzed (Participants) | 6 | 7 | 9 | 7 | 7 | 7 | 8 | 8 | 59
Age Continuous [Mean (Standard Deviation); unit: years] | 8.83 (1.33) | 9.57 (1.13) | 9.89 (1.27) | 9.71 (0.95) | 15.00 (1.83) | 13.14 (1.46) | 14.25 (1.67) | 14.00 (1.60) | 11.86 (2.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 4 | 4 | 3 | 3 | 5 | 29
  Male | 2 | 4 | 6 | 3 | 3 | 4 | 5 | 3 | 30
Children's Depression Ratings Scale-Revised (CDRS-R) total score [Mean (Standard Deviation); unit: scores on a scale] — CDRS-R total score: scale measures 17 depressive symptoms, of which 3 are rated 1 to 5 and 14 are rated 1 to 7 (1 = no symptom difficulties; 5 or 7 = severe clinically significant difficulties) for a total score range of 17 to 113. Lower total scores indicate lower intensity of symptoms.
  scores on a scale | 57.50 (4.89) | 52.43 (5.13) | 49.89 (7.30) | 46.43 (4.35) | 64.86 (11.87) | 57.71 (1.98) | 57.88 (9.19) | 48.63 (6.25) | 54.17 (8.78)

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Change From Baseline in Children's Depression Ratings Scale-Revised (CDRS-R) Total Score
Description: CDRS-R total score: scale measures 17 depressive symptoms, of which 3 are rated 1 to 5 and 14 are rated 1 to 7 (1 = no symptom difficulties; 5 or 7 = severe clinically significant difficulties) for a total score range of 17 to 113. Lower total scores indicate lower intensity of symptoms.
Time Frame: Baseline, Inpatient Days 1 to 4, Outpatient Days 5 to 7, Outpatient Weeks 2 through 8 and Outpatient Week >8 (or early termination)
Population: ITT: all treatment-assigned subjects with a baseline primary efficacy evaluation, at least 1 dose of study treatment, and at least 1 primary efficacy evaluation after the first dose of study treatment.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Desvenlafaxine 10 mg Children | Desvenlafaxine 25 mg Children | Desvenlafaxine 50 mg Children | Desvenlafaxine 100 mg Children | Desvenlafaxine 25 mg Adolescent | Desvenlafaxine 50 mg Adolescent | Desvenlafaxine 100 mg Adolescent | Desvenlafaxine 200 mg Adolescent
Number analyzed (Participants) | 6 | 7 | 9 | 7 | 7 | 7 | 8 | 8
scores on a scale
  Inpatient Days 1 to 4 | -6.83 (6.15) | -9.86 (5.40) | -2.78 (3.07) | -6.43 (10.00) | -7.00 (18.18) | -4.57 (2.99) | -8.25 (4.33) | -10.38 (13.45)
  Outpatient Days 5 to 7 | -10.67 (6.44) | -13.86 (8.51) | -10.44 (10.79) | -7.86 (8.28) | -8.00 (13.88) | -8.29 (4.27) | -9.50 (8.11) | -11.25 (14.00)
  Outpatient Week 2 | -17.67 (6.92) | -18.86 (10.51) | -14.44 (12.68) | -9.57 (10.83) | -8.29 (13.46) | -11.29 (5.53) | -18.13 (11.12) | -13.13 (14.88)
  Outpatient Week 3 | -19.67 (6.77) | -18.57 (7.93) | -16.89 (13.49) | -10.43 (9.11) | -11.71 (13.23) | -14.57 (6.19) | -21.25 (10.99) | -13.13 (11.47)
  Outpatient Week 4 | -19.50 (6.50) | -20.86 (10.98) | -17.56 (15.99) | -10.00 (4.69) | -14.57 (14.06) | -19.43 (9.43) | -23.50 (10.69) | -12.50 (9.41)
  Outpatient Week 5 | -19.50 (6.50) | -23.00 (8.56) | -19.56 (13.46) | -10.29 (4.39) | -14.57 (14.06) | -19.43 (9.43) | -23.88 (10.36) | -12.50 (9.41)
  Outpatient Week 6 | -21.83 (6.77) | -19.86 (9.94) | -18.44 (13.79) | -12.00 (5.48) | -20.57 (18.98) | -17.14 (6.20) | -24.63 (8.99) | -14.38 (9.93)
  Outpatient Week 7 | -21.83 (6.77) | -20.43 (10.06) | -19.11 (13.20) | -12.00 (5.48) | -20.57 (18.98) | -17.14 (6.20) | -25.38 (7.87) | -14.50 (9.89)
  Outpatient Week 8 | -22.00 (7.01) | -20.29 (7.18) | -19.78 (14.49) | -14.14 (6.52) | -21.43 (19.86) | -22.29 (3.09) | -27.25 (6.78) | -15.38 (8.65)
  Outpatient Week >8 | -22.00 (7.01) | -20.00 (7.05) | -19.89 (14.51) | -14.14 (6.52) | -21.43 (19.86) | -22.29 (3.09) | -26.75 (7.42) | -15.38 (8.65)

2. Other Pre Specified Outcome: Change From Baseline in Hamilton Rating Scale for Depression 17-item (HAMD-D17) Total Score
Description: HAM-D, clinician-rated interview, measures presence of depressive symptoms in 17 areas (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, & weight loss). Total score ranges from 0 to 52; higher scores reflect higher severity of current illness states.
Time Frame: as for outcome 1
Population: ITT
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Desvenlafaxine 10 mg Children | Desvenlafaxine 25 mg Children | Desvenlafaxine 50 mg Children | Desvenlafaxine 100 mg Children | Desvenlafaxine 25 mg Adolescent | Desvenlafaxine 50 mg Adolescent | Desvenlafaxine 100 mg Adolescent | Desvenlafaxine 200 mg Adolescent
Number analyzed (Participants) | 6 | 7 | 9 | 7 | 7 | 7 | 8 | 8
Score on a scale
  Inpatient Days 1 to 4 | -6.00 (5.73) | -5.43 (4.31) | -0.33 (1.94) | -2.43 (6.92) | -2.29 (7.45) | -0.57 (1.13) | -1.50 (4.54) | -5.63 (7.42)
  Outpatient Days 5 to 7 | -6.00 (5.73) | -5.43 (4.31) | -0.33 (1.94) | -2.43 (6.92) | -2.00 (7.59) | -0.57 (1.13) | -1.50 (4.54) | -5.63 (7.42)
  Outpatient Week 2 | -9.33 (7.00) | -10.71 (4.61) | -6.11 (2.67) | -5.57 (4.20) | -2.71 (4.27) | -5.71 (3.40) | -8.13 (4.91) | -9.38 (7.41)
  Outpatient Week 3 | -9.33 (7.00) | -10.29 (5.41) | -6.11 (2.67) | -5.57 (4.20) | -2.71 (4.27) | -5.71 (3.40) | -8.13 (4.91) | -8.88 (6.33)
  Outpatient Week 4 | -11.00 (5.62) | -13.00 (6.30) | -7.22 (5.61) | -7.57 (3.05) | -7.29 (5.19) | -7.57 (2.99) | -12.13 (5.69) | -9.00 (5.24)
  Outpatient Week 5 | -11.00 (5.62) | -14.14 (4.10) | -7.56 (5.64) | -9.00 (1.91) | -7.29 (5.19) | -7.57 (2.99) | -12.25 (5.73) | -9.00 (5.24)
  Outpatient Week 8 | -12.17 (6.01) | -14.00 (4.62) | -8.44 (6.88) | -11.14 (4.14) | -11.14 (9.56) | -9.86 (3.93) | -14.25 (3.96) | -11.63 (5.40)
  Outpatient Week >8 | -12.17 (6.01) | -13.86 (4.81) | -9.11 (6.68) | -11.14 (4.14) | -11.14 (9.56) | -9.86 (3.93) | -13.00 (5.37) | -11.63 (5.40)

3. Other Pre Specified Outcome: Percentage of Participants With a Categorical Clinical Global Impressions Scale-Severity (CGI-S) Score at Every Visit
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1=normal, not ill at all, 2=borderline mentally ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, 7=among the most extremely ill patients. Higher scores reflect higher severity of current illness states.
Time Frame: as for outcome 1
Population: ITT; no participants had a CGI-S score of 6 or 7, therefore only scores 1 through 5 are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Desvenlafaxine 10 mg Children | Desvenlafaxine 25 mg Children | Desvenlafaxine 50 mg Children | Desvenlafaxine 100 mg Children | Desvenlafaxine 25 mg Adolescent | Desvenlafaxine 50 mg Adolescent | Desvenlafaxine 100 mg Adolescent | Desvenlafaxine 200 mg Adolescent
Number analyzed (Participants) | 6 | 7 | 9 | 7 | 7 | 7 | 8 | 8
percentage of participants
  Inpatient Days 1 to 4: not ill at all | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Inpatient Days 1 to 4: borderline ill | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Inpatient Days 1 to 4: mildly ill | 0.0 | 0.0 | 0.0 | 14.3 | 0.0 | 0.0 | 0.0 | 12.5
  Inpatient Days 1 to 4: moderately ill | 100 | 100 | 88.9 | 85.7 | 100 | 100 | 100 | 87.5
  Inpatient Days 1 to 4: markedly ill | 0.0 | 0.0 | 11.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Days 5 to 7: not ill at all | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Days 5 to 7: borderline ill | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Days 5 to 7: mildly ill | 0.0 | 42.9 | 44.4 | 0.0 | 0.0 | 14.3 | 0.0 | 12.5
  Outpatient Days 5 to 7: moderately ill | 100 | 57.1 | 55.6 | 100 | 100 | 85.7 | 100 | 87.5
  Outpatient Days 5 to 7: markedly ill | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 2: not ill at all | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 2: borderline ill | 0.0 | 14.3 | 11.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 2: mildly ill | 66.7 | 57.1 | 55.6 | 0.0 | 0.0 | 28.6 | 50 | 12.5
  Outpatient Week 2: moderately ill | 33.3 | 28.6 | 33.3 | 100 | 100 | 71.4 | 50 | 87.5
  Outpatient Week 2: markedly ill | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 3: not ill at all | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 3: borderline ill | 0.0 | 57.1 | 0.0 | 0.0 | 0.0 | 0.0 | 25 | 0.0
  Outpatient Week 3: mildly ill | 66.7 | 42.9 | 88.9 | 0.0 | 28.6 | 57.1 | 37.5 | 12.5
  Outpatient Week 3: moderately ill | 33.3 | 0.0 | 11.1 | 100 | 71.4 | 42.9 | 37.5 | 87.5
  Outpatient Week 3: markedly ill | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 4: not ill at all | 0.0 | 14.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 4: borderline ill | 16.7 | 57.1 | 11.1 | 0.0 | 0.0 | 0.0 | 50 | 0.0
  Outpatient Week 4: mildly ill | 66.7 | 28.6 | 66.7 | 14.3 | 28.6 | 85.7 | 12.5 | 37.5
  Outpatient Week 4: moderately ill | 16.7 | 0.0 | 22.2 | 85.7 | 71.4 | 14.3 | 37.5 | 62.5
  Outpatient Week 4: markedly ill | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 5: not ill at all | 0.0 | 14.3 | 11.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 5: borderline ill | 16.7 | 57.1 | 11.1 | 0.0 | 0.0 | 0.0 | 50 | 0.0
  Outpatient Week 5: mildly ill | 66.7 | 28.6 | 55.6 | 14.3 | 28.6 | 85.7 | 12.5 | 37.5
  Outpatient Week 5: moderately ill | 16.7 | 0.0 | 22.2 | 85.7 | 71.4 | 14.3 | 37.5 | 62.5
  Outpatient Week 5: markedly ill | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 6: not ill at all | 0.0 | 0.0 | 11.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 6: borderline ill | 50 | 57.1 | 11.1 | 0.0 | 0.0 | 14.3 | 62.5 | 0.0
  Outpatient Week 6: mildly ill | 50 | 42.9 | 66.7 | 28.6 | 57.1 | 57.1 | 12.5 | 50
  Outpatient Week 6: moderately ill | 0.0 | 0.0 | 11.1 | 71.4 | 42.9 | 28.6 | 25 | 50
  Outpatient Week 6: markedly ill | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 7: not ill at all | 0.0 | 0.0 | 11.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 7: borderline ill | 50 | 42.9 | 11.1 | 0.0 | 0.0 | 14.3 | 62.5 | 0.0
  Outpatient Week 7: mildly ill | 50 | 57.1 | 77.8 | 28.6 | 57.1 | 57.1 | 25 | 50
  Outpatient Week 7: moderately ill | 0.0 | 0.0 | 0.0 | 71.4 | 42.9 | 28.6 | 12.5 | 50
  Outpatient Week 7: markedly ill | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 8: not ill at all | 0.0 | 0.0 | 11.1 | 0.0 | 0.0 | 0.0 | 12.5 | 0.0
  Outpatient Week 8: borderline ill | 66.7 | 42.9 | 22.2 | 0.0 | 0.0 | 28.6 | 50 | 0.0
  Outpatient Week 8: mildly ill | 33.3 | 57.1 | 66.7 | 71.4 | 57.1 | 71.4 | 25 | 62.5
  Outpatient Week 8: moderately ill | 0.0 | 0.0 | 0.0 | 28.6 | 42.9 | 0.0 | 12.5 | 37.5
  Outpatient Week 8: markedly ill | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week >8: not ill at all | 0.0 | 0.0 | 11.1 | 0.0 | 0.0 | 0.0 | 12.5 | 0.0
  Outpatient Week >8: borderline ill | 66.7 | 57.1 | 33.3 | 0.0 | 0.0 | 28.6 | 50 | 0.0
  Outpatient Week >8: mildly ill | 33.3 | 42.9 | 55.6 | 71.4 | 57.1 | 71.4 | 25 | 62.5
  Outpatient Week >8: moderately ill | 0.0 | 0.0 | 0.0 | 28.6 | 42.9 | 0.0 | 12.5 | 37.5
  Outpatient Week >8: markedly ill | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

4. Primary Outcome: Number of Participants With Adverse Events AEs) and Serious Adverse Events (SAEs)
Description: AEs are any untoward, undesired, or unplanned event in the form of signs, symptoms, disease, or laboratory or physiologic observations occurring in a person given study treatment. The event does not need to be causally related to the study treatment. SAEs are adverse events that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in persistent or significant disability or incapacity, result in cancer, or result in a congenital anomaly or birth defect.
Time Frame: Baseline to Follow-up (up to Day 77)
Population: Safety population includes all treatment-assigned participants who have taken at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Desvenlafaxine 10 mg Children | Desvenlafaxine 25 mg Children | Desvenlafaxine 50 mg Children | Desvenlafaxine 100 mg Children | Desvenlafaxine 25 mg Adolescent | Desvenlafaxine 50 mg Adolescent | Desvenlafaxine 100 mg Adolescent | Desvenlafaxine 200 mg Adolescent
Number analyzed (Participants) | 6 | 7 | 9 | 7 | 7 | 7 | 8 | 8
participants
  Serious Adverse Events | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Non-serious Adverse Events | 1 | 3 | 3 | 7 | 4 | 2 | 7 | 8

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Noncompartmental pharmacokinetic (PK) parameter obtained using 0 to 72 hour concentration data from venous blood samples measured as nanograms per milliliter (ng/mL).
Time Frame: Pre-dose (0 hour) and Post-dose (0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours) on Days 28 and 56
Population: PK population: all participants in the Safety population with available plasma concentration data from both the inpatient and outpatient phases of the study that are properly identified with respect to dosing and sampling times.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Desvenlafaxine 10 mg Children | Desvenlafaxine 25 mg Children | Desvenlafaxine 50 mg Children | Desvenlafaxine 100 mg Children | Desvenlafaxine 25 mg Adolescent | Desvenlafaxine 50 mg Adolescent | Desvenlafaxine 100 mg Adolescent | Desvenlafaxine 200 mg Adolescent
Number analyzed (Participants) | 6 | 7 | 9 | 7 | 7 | 7 | 8 | 8
ng/mL | 33.9 (12.1) | 98 (60.5) | 108 (27) | 263 (66) | 46.1 (15.9) | 93.9 (15.5) | 202 (92) | 449 (126)

6. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: Noncompartmental PK parameter obtained using 0 to 72 hour concentration data from venous blood samples measured as hours (hr).
Time Frame: Pre-dose (0 hour) and Post-dose (0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours) on Days 28 and 56
Population: PK population
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Desvenlafaxine 10 mg Children | Desvenlafaxine 25 mg Children | Desvenlafaxine 50 mg Children | Desvenlafaxine 100 mg Children | Desvenlafaxine 25 mg Adolescent | Desvenlafaxine 50 mg Adolescent | Desvenlafaxine 100 mg Adolescent | Desvenlafaxine 200 mg Adolescent
Number analyzed (Participants) | 6 | 7 | 9 | 7 | 7 | 7 | 8 | 8
hr | 4.7 (2.1) | 4.3 (1.4) | 5.1 (3) | 5.0 (2.0) | 4.3 (0.7) | 8.7 (7.1) | 7.6 (3.4) | 7.5 (4.1)

7. Primary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Noncompartmental PK parameter obtained using 0 to 72 hour concentration data from venous blood samples measured as hours (hr).
Time Frame: Pre-dose (0 hour) and Post-dose (0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours) on Days 28 and 56
Population: PK population
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Desvenlafaxine 10 mg Children | Desvenlafaxine 25 mg Children | Desvenlafaxine 50 mg Children | Desvenlafaxine 100 mg Children | Desvenlafaxine 25 mg Adolescent | Desvenlafaxine 50 mg Adolescent | Desvenlafaxine 100 mg Adolescent | Desvenlafaxine 200 mg Adolescent
Number analyzed (Participants) | 6 | 7 | 9 | 7 | 7 | 7 | 8 | 8
hr | 7.8 (1.4) | 8.6 (1.6) | 9.4 (2.7) | 9.0 (2.0) | 12 (3) | 10.2 (3.7) | 9.6 (2.0) | 9.8 (2.7)

8. Primary Outcome: Area Under the Curve From Time Zero to Infinity (AUC0-∞)
Description: AUC (0-∞) = Area under the plasma concentration versus time curve from time zero (pre-dose) to infinity. Noncompartmental PK parameter obtained using 0 to 72 hour concentration data from venous blood samples measured as nanograms multiplied by hours divided by milliliters (ng*hr/mL).
Time Frame: Pre-dose (0 hour) and Post-dose (0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours) on Days 28 and 56
Population: PK population
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Desvenlafaxine 10 mg Children | Desvenlafaxine 25 mg Children | Desvenlafaxine 50 mg Children | Desvenlafaxine 100 mg Children | Desvenlafaxine 25 mg Adolescent | Desvenlafaxine 50 mg Adolescent | Desvenlafaxine 100 mg Adolescent | Desvenlafaxine 200 mg Adolescent
Number analyzed (Participants) | 6 | 7 | 8 | 7 | 7 | 7 | 8 | 8
ng*hr/mL | 628 (346) | 1704 (553) | 2414 (924) | 6732 (3031) | 1123 (361) | 2281 (689) | 5290 (2188) | 11730 (3113)

9. Secondary Outcome: Population Pharmacokinetics Dose Normalized AUC (AUC/D): First Method, Second Method
Description: Relationship of variables (i.e., age, sex, ethnicity, and food) examined by fitting dose normalized AUC (AUC/D) values to a power model. AUC/D regressed against variables using power equation Y=A*W^b (Y=AUC/D; A=coefficient; W=variable; b=exponent). AUC values from children cohort (ages 7 to 11) combined doses=first method of analysis. AUC from adolescent cohort (ages 12 to 17) combined doses=second method of analysis. AUC values combined from both cohorts=third method of analysis. Measured as nanograms multiplied by hours divided by milliliters per milligram of dose [(ng*hr/mL)/mg of dose].
Time Frame: Day 1, Day 28, and Day 56
Population: PK population; data was insufficient examine the effect of age, sex, ethnicity, and food on the PK of desvenlafaxine. Coefficient and exponent values were calculated for variable of body weight, however, the AUC/D values were not summarized as descriptive statistics.
Measure: Number; unit: (ng*hr/mL)/mg of dose
Groups:
- Desvenlafaxine - Combined Children Cohorts: Desvenlafaxine sustained release tablets for 10 mg, 25 mg, 50 mg, and 100 mg Children cohort dose levels.
- Desvenlafaxine - Combined Adolescent Cohorts: Desvenlafaxine sustained release tablets for 25 mg, 50 mg, 100 mg, and 200 mg Adolescent cohort dose levels.
Arm/Group | Desvenlafaxine - Combined Children Cohorts | Desvenlafaxine - Combined Adolescent Cohorts
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Population Pharmacokinetics Dose Normalized AUC (AUC/D): Third Method
Description: as for outcome 9
Time Frame: Day 1, Day 28, and Day 56
Population: as for outcome 9
Measure: Number; unit: (ng*hr/mL)/mg of dose
Groups:
- Desvenlafaxine - Combined Children and Adolescent Cohorts: Desvenlafaxine sustained release tablets for 10 mg, 25 mg, 50 mg, and 100 mg Children cohort dose levels and Desvenlafaxine sustained release tablets for 25 mg, 50 mg, 100 mg, and 200 mg Adolescent cohort dose levels.
Arm/Group | Desvenlafaxine - Combined Children and Adolescent Cohorts
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Percentage of Participants With a Categorical Clinical Global Impressions Scale-Improvement(CGI-I) Score at Every Visit
Description: CGI-I: 7-point clinician rated scale ranging from 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, to 7=very much worse. Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Scores above 4 reflect worsening of illness state as compared to baseline.
Time Frame: as for outcome 1
Population: ITT; no participants had a CGI-I score of 6 or 7, therefore only scores 1 through 5 are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Desvenlafaxine 10 mg Children | Desvenlafaxine 25 mg Children | Desvenlafaxine 50 mg Children | Desvenlafaxine 100 mg Children | Desvenlafaxine 25 mg Adolescent | Desvenlafaxine 50 mg Adolescent | Desvenlafaxine 100 mg Adolescent | Desvenlafaxine 200 mg Adolescent
Number analyzed (Participants) | 6 | 7 | 9 | 7 | 7 | 7 | 8 | 8
percentage of participants
  Inpatient Days 1 to 4: very much improved | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Inpatient Days 1 to 4: much improved | 0.0 | 0.0 | 0.0 | 14.3 | 14.3 | 0.0 | 0.0 | 12.5
  Inpatient Days 1 to 4: minimally improved | 0.0 | 0.0 | 11.1 | 0.0 | 0.00 | 0.0 | 12.5 | 37.5
  Inpatient Days 1 to 4: no change | 100 | 100 | 88.9 | 85.7 | 85.7 | 100 | 87.5 | 50
  Inpatient Days 1 to 4: minimally worse | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Days 5 to 7: very much improved | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Days 5 to 7: much improved | 0.0 | 14.3 | 11.1 | 0.0 | 0.0 | 0.0 | 0.0 | 12.5
  Outpatient Days 5 to 7: minimally improved | 50 | 14.3 | 55.6 | 42.9 | 42.9 | 57.1 | 25 | 25
  Outpatient Days 5 to 7: no change | 50 | 71.4 | 33.3 | 57.1 | 57.1 | 42.9 | 75 | 62.5
  Outpatient Days 5 to 7: minimally worse | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 2: very much improved | 0.0 | 0.0 | 11.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 2: much improved | 33.3 | 28.6 | 44.4 | 14.3 | 0.0 | 0.0 | 0.0 | 25
  Outpatient Week 2: minimally improved | 50 | 42.9 | 11.1 | 42.9 | 42.9 | 57.1 | 75 | 50
  Outpatient Week 2: no change | 16.7 | 28.6 | 33.3 | 42.9 | 57.1 | 42.9 | 25 | 25
  Outpatient Week 2: minimally worse | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 3: very much improved | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 3: much improved | 50 | 85.7 | 44.4 | 14.3 | 28.6 | 0.0 | 37.5 | 25
  Outpatient Week 3: minimally improved | 50 | 14.3 | 44.4 | 57.1 | 57.1 | 71.4 | 37.5 | 62.5
  Outpatient Week 3: no change | 0.0 | 0.0 | 11.1 | 28.6 | 14.3 | 28.6 | 25 | 12.5
  Outpatient Week 3: minimally worse | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 4: very much improved | 0.0 | 14.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 4: much improved | 50 | 71.4 | 55.6 | 28.6 | 28.6 | 0.0 | 50 | 37.5
  Outpatient Week 4: minimally improved | 50 | 14.3 | 22.2 | 57.1 | 57.1 | 85.7 | 37.5 | 37.5
  Outpatient Week 4: no change | 0.0 | 0.0 | 11.1 | 14.3 | 14.3 | 14.3 | 12.5 | 12.5
  Outpatient Week 4: minimally worse | 0.0 | 0.0 | 11.1 | 0.0 | 0.0 | 0.0 | 0.0 | 12.5
  Outpatient Week 5: very much improved | 0.0 | 14.3 | 11.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 5: much improved | 50 | 85.7 | 55.6 | 28.6 | 28.6 | 0.0 | 50 | 37.5
  Outpatient Week 5: minimally improved | 50 | 0.0 | 22.2 | 71.4 | 57.1 | 85.7 | 37.5 | 37.5
  Outpatient Week 5: no change | 0.0 | 0.0 | 0.0 | 0.0 | 14.3 | 14.3 | 12.5 | 12.5
  Outpatient Week 5: minimally worse | 0.0 | 0.0 | 11.1 | 0.0 | 0.0 | 0.0 | 0.0 | 12.5
  Outpatient Week 6: very much improved | 0.0 | 14.3 | 11.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 6: much improved | 50 | 57.1 | 66.7 | 28.6 | 57.1 | 71.4 | 75 | 50
  Outpatient Week 6: minimally improved | 50 | 28.6 | 22.2 | 71.4 | 28.6 | 28.6 | 12.5 | 25
  Outpatient Week 6: no change | 0.0 | 0.0 | 0.0 | 0.0 | 14.3 | 0.0 | 12.5 | 25
  Outpatient Week 6: minimally worse | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 7: very much improved | 0.0 | 14.3 | 11.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 7: much improved | 50 | 42.9 | 55.6 | 28.6 | 57.1 | 71.4 | 75 | 50
  Outpatient Week 7: minimally improved | 50 | 42.9 | 33.3 | 71.4 | 28.6 | 28.6 | 12.5 | 37.5
  Outpatient Week 7: no change | 0.0 | 0.0 | 0.0 | 0.0 | 14.3 | 0.0 | 12.5 | 12.5
  Outpatient Week 7: minimally worse | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week 8: very much improved | 0.0 | 14.3 | 22.2 | 0.0 | 0.0 | 0.0 | 12.5 | 0.0
  Outpatient Week 8: much improved | 83.3 | 71.4 | 22.2 | 71.4 | 57.1 | 71.4 | 75 | 62.5
  Outpatient Week 8: minimally improved | 16.7 | 14.3 | 55.6 | 28.6 | 28.6 | 28.6 | 0.0 | 37.5
  Outpatient Week 8: no change | 0.0 | 0.0 | 0.0 | 0.0 | 14.3 | 0.0 | 12.5 | 0.0
  Outpatient Week 8: minimally worse | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Outpatient Week >8: very much improved | 0.0 | 14.3 | 22.2 | 0.0 | 0.0 | 0.0 | 12.5 | 0.0
  Outpatient Week >8: much improved | 83.3 | 71.4 | 33.3 | 71.4 | 57.1 | 71.4 | 75 | 62.5
  Outpatient Week >8: minimally improved | 16.7 | 14.3 | 44.4 | 28.6 | 28.6 | 28.6 | 0.0 | 37.5
  Outpatient Week >8: no change | 0.0 | 0.0 | 0.0 | 0.0 | 14.3 | 0.0 | 12.5 | 0.0
  Outpatient Week >8: minimally worse | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Description: An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Desvenlafaxine 10 mg Children | Desvenlafaxine 25 mg Children | Desvenlafaxine 50 mg Children | Desvenlafaxine 100 mg Children | Desvenlafaxine 25 mg Adolescent | Desvenlafaxine 50 mg Adolescent | Desvenlafaxine 100 mg Adolescent | Desvenlafaxine 200 mg Adolescent
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/9 | 0/7 | 1/7 | 0/7 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/6 | 3/7 | 3/9 | 7/7 | 4/7 | 2/7 | 7/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Desvenlafaxine 10 mg Children (N=6) | Desvenlafaxine 25 mg Children (N=7) | Desvenlafaxine 50 mg Children (N=9) | Desvenlafaxine 100 mg Children (N=7) | Desvenlafaxine 25 mg Adolescent (N=7) | Desvenlafaxine 50 mg Adolescent (N=7) | Desvenlafaxine 100 mg Adolescent (N=8) | Desvenlafaxine 200 mg Adolescent (N=8)
Suicidal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Desvenlafaxine 10 mg Children (N=6) | Desvenlafaxine 25 mg Children (N=7) | Desvenlafaxine 50 mg Children (N=9) | Desvenlafaxine 100 mg Children (N=7) | Desvenlafaxine 25 mg Adolescent (N=7) | Desvenlafaxine 50 mg Adolescent (N=7) | Desvenlafaxine 100 mg Adolescent (N=8) | Desvenlafaxine 200 mg Adolescent (N=8)
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 2 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 5
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Application site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling jittery (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 3 | 1 | 1 | 2 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 4
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Affect lability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.